CLINICAL TRIAL: NCT04109859
Title: Effect of Methylene Blue on Perioperative Organ Function in Patients With Obstructive Jaundice
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Jiaolin Ning,MD (Other)
Responsible Party: Sponsor-Investigator, Jiaolin Ning,MD, Professor of department of anesthesia, Southwest Hospital, China
Organization: Southwest Hospital, China (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY201999
Record Dates: First submitted 2019-09-25; First posted 2019-09-30 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Jaundice
MeSH Terms: conditions — Jaundice | interventions — Sodium Chloride; Methylene Blue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Methylene blue group (Experimental): Before the anesthesia was intubated, the patients in the methylene blue group were given a 2 mg/Kg methylene blue 50 ml intravenously for 10 min; continuous constant speed pumping methylene blue(0.5mg/Kg/h).
  Interventions: Drug: Methylene Blue
- Placebo group (Placebo Comparator): Before the anesthesia was intubated, the placebo group was given 50 ml of normal saline for 10 min.continuous constant speed pumpingnormal saline (10ml/h).
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Saline — When using saline, if found mean arterial pressure <65mmHg, Cardic Output>4L/min, Sequential Vascular Response<800 (dyne×sec)/cm, starting dose of norepinephrine 0.04ug/min/kg
  Other Names: Placebo group
  Arms: Placebo group
Drug: Methylene Blue — Patients in the methylene blue group were given methylene blue before anesthesia and continued intraoperative pumping
  Other Names: Methylene blue group
  Arms: Methylene blue group

SUMMARY:
Increased production of vasodilating substances such as NO plays an important role in the development of vasoplegic syndrome caused by obstructive jaundice.Methylene blue plays a role in raising blood pressure by inhibiting the vasodilator Nitric Oxide (NO)

DETAILED DESCRIPTION:
The level of circulating hydrogen sulfide (H2S) in patients with obstructive jaundice is significantly increased. As a direct opener of KATP channels in vivo, H2S also has diastolic peripheral vasculature . H2S participates in the occurrence of vasoplegic syndrome in patients with obstructive jaundice by interacting with NO. However, it is unclear whether methylene blue can relieve vasoplegic syndrome in patients with obstructive jaundice by inhibiting the vasodilating effect of substances such as H2S and NO.

Therefore, this clinical study intends to include patients with obstructive jaundice, using randomized, controlled, prospective study to explore the effect of methylene blue on the occurrence of vasoplegic syndrome, organ function and prognosis in patients with obstructive jaundice.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18~70 years old;
2. ASA grade I~III;
3. Ability to comply with research protocols;
4. Patients with obstructive jaundice: patients with total bilirubin greater than 50umol/L;
5. Voluntarily participate in the study and sign the informed consent form. -

Exclusion Criteria:

1. ASA IV~V grade;
2. women during lactation and pregnancy;
3. Patients with severe heart disease or lung disease before surgery;
4. Participating in other trials in the last 2 months;
5. Those whose mental state cannot cooperate, who suffer from mental illness, have no self-control, and cannot express clearly;
6. Those who refuse to sign the informed consent form. -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-01-21 (Estimated); Study Completion 2021-01-21 (Estimated)

PRIMARY OUTCOMES:
Acute physiology and chronic health evaluation IIScore sheet | 3 days
  use this Score sheet to evaluation of postoperative organ function in patients.The total score is 0 to 71

CONTACTS AND LOCATIONS:
Overall Officials: Jiaolin Ning, MD, Principal Investigator — Professor of department of anesthesia, Southwest Hospital
Locations (1):
- department of anesthesia, Southwest Hospital, Third Military Medical University Affiliation: Southwest Hospital, China, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No